CLINICAL TRIAL: NCT07063602
Title: Sensory Anesthesia Achieved Through Different Paravertebral Block Approaches for Post-Operative Pain Management After Videothoracoscopic Lung Resection
Brief Title: Sensory Anesthesia Achieved Through Different Paravertebral Block Approaches for Post-Op Pain Management After VATS Lung Resection
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2026-13022
Record Dates: First submitted 2025-06-30; First posted 2025-07-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Thoracic Surgery; Video-assisted; Paravertebral Block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paravertebral block using the percutaneous or the transpleural technique: The investigators aim to conduct a prospective observational study including patients having a paravertebral block undergoing a VATS lung surgery. The paravertebral block administration technique will vary sequentially, meaning that the first 30 patients included will receive the percutaneous technique, and the next 30 will receive the transpleural technique.
  Paravertebral block will be administered at two levels, T4 and T7, using the percutaneous or the transpleural technique. It will be administered by the surgeon directly after the installation of the thoracoscope and before the start of lung and lymph node resection. The local anesthetic will be bupivacaine 0.5% with 5 mcg/mL of adrenaline for a total volume of 0.4 mL/kg.
  Interventions: Other: Evaluation of the hypoesthesia of the thorax

INTERVENTIONS:
Other: Evaluation of the hypoesthesia of the thorax — In the recovery room, a member of the research team will come to assess the presence of hypoesthesia (loss of sensation) of the thorax using ice and a Von Frey filament applied at three different sections: midscapular, midaxillary and midclavicular.

SUMMARY:
Video-assisted thoracoscopic lung resection (VATS) is a minimally invasive surgical approach frequently used in the treatment of lung cancers. The most commonly used analgesic technique for this surgery is the paravertebral block with a single peroperative injection of local anesthetic. However, a recent study conducted at our institution revealed that this approach provided less relief than expected in some patients. In light of these results, it becomes crucial to distinguish between technical failures (absence of sensitive anesthesia) and the intrinsic limits of the chosen regional analgesia technique (pain originating from an unanesthetized area or pain despite the presence of sensitive anesthesia) in order to better relieve patients.

This study aims to objectively assess the areas of anesthesia obtained through two methods of paravertebral block to evaluate their respective performance and optimize post-VATS analgesic management.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic lung resection (VATS) is a minimally invasive surgical approach frequently used in the treatment of lung cancers. Compared to traditional thoracotomy, it is associated with reduced acute postoperative pain and a faster recovery. However, this pain often remains moderate to severe and can, if poorly controlled, promote the development of chronic pain. A multimodal analgesic strategy is essential to limit the use of opioids and their side effects. The most commonly used analgesic technique is the paravertebral block. As part of the optimized recovery protocols at our institution, a single peroperative injection of local anesthetic, guided by thoracoscopy, is currently favored. This technique, which is simple and safe, promotes rapid mobilization of the patient. However, a recent study conducted at our institution revealed that this approach provided less relief than expected in some patients. In light of these results, it becomes crucial to distinguish between technical failures (absence of sensitive anesthesia) and the intrinsic limits of the chosen regional analgesia technique (pain originating from an unanesthetized area or pain despite the presence of sensitive anesthesia) in order to better relieve patients.

This study aims to objectively assess the areas of anesthesia obtained through two methods of paravertebral block to evaluate their respective performance and optimize post-VATS analgesic management.

The primary objective of the study is to compare the success rate of creating sensitive anesthesia of the thoracic wall in the acute postoperative phase of video-assisted thoracoscopic lung resection according to various administration methods (transpleural vs percutaneous approach).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* American Society of Anesthesiologists (ASA) score 1-3

Exclusion Criteria:

* Contraindication to the paravertebral block (coagulopathy, use of anticoagulants or antiplatelet agents other than aspirin that have not been stopped according to hospital guidelines, thoracoscopic visualization of the paravertebral space expected to be difficult or impossible, anterior spinal surgery with potential discontinuity of the paravertebral space)
* Epidural analgesia preferred (high risk of thoracotomy, marginal lung function)
* Surgical criteria: conversion to thoracotomy necessary and thoracic epidural or other form of regional analgesia implemented post-operatively
* Known allergy to local anesthetics
* Language barrier, psychiatric, physical or mental condition making pain assessment impossible despite prior education
* Pregnancy
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective anatomical pulmonary resection by VATS at our institution
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Success rate of the sensory block | One hour after the surgery
  The success rate of the sensory block, defined as a hypoesthetic level to ice or the Von Frey filament of at least T3 to T8 in the recovery room, assessed at mid-scapular, mid-axillary, and mid-clavicular.

SECONDARY OUTCOMES:
Severity of acute postoperative pain | One hour after the surgery
  The severity of acute postoperative pain according to the visual analog scale for pain (VAS, 0 to 100 mm, where 0 means "no pain" and 100 means the "worst possible pain.") at rest and during coughing, at the thorax 1 hour after surgery.
Postoperative morphine-equivalents consumption | Perioperative
  The total amount of morphine equivalents received perioperatively, including pre-emergence and recovery room doses.
Total duration in the operating room | At the end of the surgery
  Total lenght of stay of the patient in the operating room
Time to recovery room discharge | 24 hours
  The time before reaching the discharge criteria for the patient to leave the recovery room
Quality of the local anesthetic diffusion | After the parabertebral block, during the surgery
  The anesthesiologist in the operating room or the surgeon will visually assess the quality of local anesthetic diffusion (approximate number of levels) following the paravertebral block, considering possible technical or anatomical constraints.
Incidence of nausea related to opioid consumption | 24 hours
  Evaluation of the incidence of nausea (yes or no) in the recovery room
Incidence of vomiting related to opioid consumption | 24 hours
  Evaluation of the incidence of vomiting (yes or no) in the recovery room
Incidence of pruritus related to opioid consumption | 24 hours
  Evaluation of the incidence of pruritus (yes or no) in the recovery room
Incidence of postoperative hypotension requiring medical intervention | 24 hours
  Evaluation of the incidence of postoperative hypotension requiring medical intervention (yes or no) in the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Alex Moore, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada